CLINICAL TRIAL: NCT03720353
Title: Pharmacological Intervention for Symptomatic Snoring
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Scott Aaron Sands, Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018P002094
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Snoring
MeSH Terms: conditions — Snoring

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active H (Active Comparator): Participants will take SAS2094AL and SAS2094BH for 3 days, then SAS2094AH and SAS2094BH for 7 days.
  Interventions: Drug: SAS2094AH and SAS2094BH
- Active L (Active Comparator): Participants will take SAS2094AL and SAS2094BL for 10 days
  Interventions: Drug: SAS2094AL and SAS2094BL
- Placebo (Placebo Comparator): Participants will take placebo for 10 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAS2094AH and SAS2094BH — SAS2094AH and SAS2094BH for 7 days, preceded by SAS2094AL and SAS2094BH for 3 days.
  Arms: Active H
Drug: SAS2094AL and SAS2094BL — SAS2094AL and SAS2094BL for 10 days
  Arms: Active L
Drug: Placebo — Placebo for 10 days. Capsules will mimic active treatments.
  Arms: Placebo

SUMMARY:
Currently, there is no pharmacological intervention capable of maintaining airway patency for the treatment of snoring and airflow limitation during sleep. Here we study the effect of pharmacological stimulation of the pharyngeal muscles on snoring severity, in a randomized quadruple-blind, crossover study.

DETAILED DESCRIPTION:
Two active interventions are being studied and compared against placebo. Participants will therefore be randomized to one of six possible sequences. Washout periods will be 1 week.

Effects of interventions on outcomes will be assessed using mixed effect model analyses: we will quantify the effect of active treatment 1 (referenced to placebo), the effect of active treatment 2 (referenced to placebo), adjusting for effects of time (period number), carryover effects, and baseline values (fixed effects). Participants are considered random effects.

Primary outcome is based on significance of active intervention 1 versus placebo.

ELIGIBILITY:
Inclusion Criteria for Enrollment

* Age 18-79 yrs
* Self-reported habitual snoring ("most of the time" or "all of the time" on Snoring Self-Evaluation Scale)
* Sleep-related symptoms defined by any of the following*:

  * Visual-Analog Scale for Sleep Quality ≤7/10 ("reduced sleep quality")
  * Epworth Sleepiness Scale ≥10 ("excessive daytime sleepiness")
  * Functional Outcomes of Sleep Questionnaire <18 ("reduced sleep-related quality of life").
* Presence of a bed-partner who is able to provide feedback to the participant on snoring (Snoring Bed-Partner Evaluation Scale)

  * The intention of these criteria is to enable participants with a broad range of possible snoring symptoms to be included. We note that the Visual-Analog Scale for Sleep Quality is, on average, approximately 7/10 in patients with sleep apnea; thus, we consider a value at or below 7 to indicate "reduced sleep quality".

Exclusion Criteria for Enrollment

* Known obstructive sleep apnea (OSA, except "mild")
* Current treatment for OSA or snoring (continuous positive airway pressure, oral appliances, supplemental oxygen)
* Use of medications expected to stimulate or depress respiration (including opioids, barbiturates, acetazolamide, doxapram, almitrine, theophylline, 4-hydroxybutanoic acid).
* Use of similar medications to the study drugs.
* Conditions likely to affect obstructive sleep apnea physiology: neuromuscular disease or other major neurological disorder, heart failure (also below), or any other unstable major medical condition.
* Respiratory disorders other than sleep disordered breathing:

  o chronic hypoventilation/hypoxemia (awake oxygen saturation < 92% by oximetry) due to chronic obstructive pulmonary disease or other respiratory conditions.
* Other sleep disorders: periodic limb movements (periodic limb movement arousal index > 10/hr), narcolepsy, or parasomnias.
* Contraindications to the study drugs, including:

  * clinically-significant kidney disorders (eGFR<60 ml/min/1.73m2)
  * clinically-significant liver disorders
  * clinically-significant cardiovascular conditions

    * severe hypertension (systolic blood pressure above 180 mmHg or diastolic below 110 mmHg measured at baseline)
    * cardiomyopathy (left ventricular ejection fraction, LVEF<50%) or heart failure
    * advanced atherosclerosis
    * history of cerebrovascular events
    * history of cardiac arrhythmias e.g., atrial fibrillation, QT prolongation
    * other serious cardiac conditions
  * myasthenia gravis
  * pregnancy/breast-feeding

We will not make new measurements of eGFR, LVEF or document their presence/absence for each participant.

Criteria for Randomization

After the baseline visit, the following criteria need to be met to continue participation:

* Participants with AHI≥15 events/hr (moderate-to-severe OSA, hypopneas based on a 30% reduction in flow, accompanied by either a 3% oxygen desaturation or scored EEG-arousal) on the baseline study night, will not continue further participation after the baseline visit.
* Participants must exhibit evidence of snoring during the baseline sleep study for further participation (mean tracheal sound intensity, Leq, exceeding 80 dB); the precise cutoff will be pilot tested in ongoing protocols (where snoring is routinely measured).

Thus, strictly, the study population will include patients with symptomatic habitual snoring, with or without mild OSA (i.e. AHI<5 and 5≤AHI<15). We note that studies in patients with moderate-to-severe OSA have already been performed (AHI>15), and further studies in this population are in progress. The inclusion of "mild OSA" will prevent a gap in the inclusion criteria for the investigation of the current intervention.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Snoring intensity | 1 week
  mean tracheal snoring sound intensity (tracheal microphone), decibels

SECONDARY OUTCOMES:
Snoring frequency | 1 week
  snoring frequency (tracheal microphone), snores per hour of total sleep time
Snoring Self-Evaluation Scale | 1 week
  frequency, loudness, disruption, bothersome, 5-point scales
Snoring Bed-Partner Evaluation Scale | 1 week
  frequency, loudness, disruption, bothersome, 5-point scales
Flow-limitation frequency | 1 week
  breaths per hour (nasal pressure airflow shape)
Flow-limitation severity | 1 week
  flow:drive ratio (nasal pressure airflow shape), %
Visual-Analog Scale for Sleep Quality | 1 week
  0-10 scale
Mean oxygen saturation | 1 week
  Percentage
Stage 1 Sleep | 1 week
  %Total sleep time
Arousal index | 1 week
  events per hour of total sleep time
Visual-Analog Scale for Treatment Satisfaction | 1 week
  0-10 scale
Epworth Sleepiness Scale | 1 week
  units on a scale
Functional Outcomes of Sleep Questionnaire | 1 week
  30 items, units on a scale
"Would you keep using this medication?" | 1 week
  Yes/No

OTHER OUTCOMES:
Maximum Tracheal Snoring Sound Intensity | 1 week
  Maximum Tracheal Snoring Sound Intensity, "L1", based on 99th percentile of snoring sound intensity expressed in decibels (dB)
Visual-Analog Scales for Excessive Fatigue | 1 week
  0-10 scale
Visual-Analog Scales for Wake-up Unrefreshed | 1 week
  0-10 scale
Visual-Analog Scales for Low Energy | 1 week
  0-10 scale

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Sands, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data will be owned by study Sponsor Apnimed, and may be made available per request.

REFERENCES:
- [Derived] Calianese N, Hess LB, Vena D, Konefal R, Mann DL, Taranto-Montemurro L, Bertisch SM, Sofer T, Azarbarzin A, Gell LK, Sands SA. Atomoxetine plus oxybutynin for symptomatic snoring and airflow limitation in individuals without moderate-to-severe obstructive sleep apnea. J Clin Sleep Med. 2025 Sep 1;21(9):1579-1590. doi: 10.5664/jcsm.11760. PMID 40471069